CLINICAL TRIAL: NCT03385993
Title: Digital Rehabilitation Environment Augmenting Medical System
Acronym: DREAMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201703107
Record Dates: First submitted 2017-12-20; First posted 2017-12-29 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Delirium
Keywords: Delirium Prevention; Virtual Reality; VR
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mediation and Relaxation Intervention (Experimental): Patients will undergo a technology based guided meditation and relaxation exercise through use of an application on a tablet or virtual reality headset.
  Interventions: Device: Technology based guided meditation and relaxation

INTERVENTIONS:
Device: Technology based guided meditation and relaxation — Subjects will be guided through a mediation and relaxation exercise on a tablet or virtual reality headset for up to an hour each day.

SUMMARY:
D.R.E.A.M.S. will assess an immersive digital reality-augmenting system in reducing the occurrence of cognitive, behavioral, and emotional consequences of critical illness and environmental exposures that are risk factors for the development of delirium.

DETAILED DESCRIPTION:
The purpose of Digital Rehabilitation Environment Augmenting Medical System (D.R.E.A.M.S.) is to research the feasibility and clinical potential of an immersive digital reality-augmenting system in reducing the occurrence of cognitive, behavioral, and emotional consequences of critical illness (e.g. pain, anxiety and insomnia) and environmental exposures (noise & light) that are risk factors for the development of delirium, a common and devastating complication in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years admitted to University of Florida (UF) Health Shands Hospital who do not have a positive Confusion Assessment Method (CAM) score, including ICU patients.

Exclusion Criteria: The study team will exclude patients if:

* Their anticipated ICU stay is less than one day
* Patient is intubated and cannot communicate.
* Age: < 18 years
* Patient with recent (within 6 months) neuro-vascular event, intra-cranial surgery, and/or acute neurological condition as primary ICU admission reason
* Baseline cognitive impairment (e.g., advanced dementia)
* Patients who are unable to wear or use the DREAMS equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of anxiety measured by Hospital Anxiety and Depression Scale (HADS) questionnaire | Immediately before and after each intervention Up to 7 days
  The assessment is used to gauge the subject's level of anxiety and depression 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Blood Pressure -Systolic | Immediately before and after each intervention up to 7 days
  Alterations to vital signs allow for Non-Verbal Pain assessments
Heart Rate | Immediately before and after each intervention up to 7 days
  Alterations to vital signs allow for Non-Verbal Pain assessments

SECONDARY OUTCOMES:
Respiratory Rate | Entire ICU stay up to 7 days
  Alterations to vital signs allow for Non-Verbal Pain assessments
Patient pain perception | Immediately before and after each intervention up to 7 days
  Defense and Veterans Pain Rating Scale (DVPRS) Likert Scale 0 - 10, with 10 = severe pain (as bad as it could be. nothing else matters)
Amount of sedatives requested by subjects | Entire ICU stay up to 7 days
  Richmond Agitation-Sedation Scale (RASS)- Patients with a RASS of -3 or less should have their sedation decreased or modified in order to achieve a RASS of -2 to 0. Patients with a RASS of 2 to 4 are not sedated enough and should be assessed for pain, anxiety, or delirium. The underlying etiology of the agitation should be investigated and appropriately treated to achieve a RASS of -2 to 0.
Amount of sedatives subjects receive | Entire ICU stay up to 7 days
  Richmond Agitation-Sedation Scale (RASS)- Patients with a RASS of -3 or less should have their sedation decreased or modified in order to achieve a RASS of -2 to 0. Patients with a RASS of 2 to 4 are not sedated enough and should be assessed for pain, anxiety, or delirium. The underlying etiology of the agitation should be investigated and appropriately treated to achieve a RASS of -2 to 0.
Subject's quality of sleep | Daily up to 14 days
  Richards-Campbell Sleep Questionnaire (RCSQ) five-item, visual analogue scale was designed as an outcome measure for assessing the perception of sleep in critically ill patients. The scale evaluates perceptions of depth of sleep, sleep onset latency, number of awakenings, time spent awake, and overall sleep quality.
DREAMS usability and acceptability questionnaire | After each intervention up to 14 days
  A qualitative assessment of the usability and efficacy of the system Likert Scale 1-5, with 5 = strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Bihorac, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No